CLINICAL TRIAL: NCT04912219
Title: Microneedling for Dermatoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Cooper-Microneedling
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Solar Purpura
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: Microneedling
- Control (No Intervention)

INTERVENTIONS:
Device: Microneedling — Skin will be pretreated with topical 15% lidocaine creaml for 20 minutes. Water-soaked gauze will then be used to remove the lidocaine gel. Treated skin will be cleaned with 70% ethyl alcohol, allowed to dry, and then treated with hyaluronic acid gel.
  Manual traction will be applied to the skin of the treatment arm, and the SkinPen microneedle device with 0.5mm microneedles attached will be passed over the forearm skin in a cross-hatch pattern until an endpoint of fine pinpoint bleeding is achieved.
  Manual pressure with sterile ice water compresses will be used until hemostasis is achieved.
  This will be repeated for a total of four treatments one month apart
  Arms: Treatment

SUMMARY:
We hypothesize that a series of treatments with a microneedling protocol will lead to increased dermal thickness as measured by biopsy, ultrasound, and skin calipometry; an improvement in dermatology-related quality of life; and a reduction in the number of ecchymoses and skin tears, of the research subjects.

DETAILED DESCRIPTION:
Dermatoporosis is a common condition, affecting between 30-37% of the population greater than age 65. It may lead to easy bruising, skin tearing, infections, and scars.

The pathogenesis of dermatoporosis involves decreased expression of collagen I, collagen III, and collagen IV; upregulation of matrix metalloproteinases 1, 2, and 3; downregulation of issue inhibitor of matrix metalloprotein I; loss of elastic tissue; defective fibroblast synthesis of collagen; and loss of hyaluronic acid.

Microneedling, also known as percutaneous collagen induction therapy, is a safe, established technique for treatment of acne scarring, rhytides, cellulite, and improvement of skin texture.

Microneedling has been demonstrated to stimulate growth factor release and increase dermal collagen and elastic fibers. It is effective in improving facial laxity, acne scarring, and facial rhytides.

Microneedling is safe and well tolerated. Expected adverse events include bleeding and oozing of the skin surface, redness, swelling, and peeling. Reported complications include post-inflammatory pigmentary changes, granulomatous reactions and systemic hypersensitivity reactions.

References:

1. Wollina U, Lotti T, Vojvotic A, Nowak A. Dermatoporosis - The Chronic Cutaneous Fragility Syndrome. Open Access Maced J Med Sci. 2019;7(18):3046-3049.
2. Dyer JM, Miller RA. Chronic Skin Fragility of Aging: Current Concepts in the Pathogenesis, Recognition, and Management of Dermatoporosis. J Clin Aesthet Dermatol. 2018;11(1):13-18.
3. McCrudden MT, McAlister E, Courtenay AJ, Gonzalez-Va ́zquez P, Singh TR, Donnelly RF Microneedle applications in improving skin appearance. Exp Dermatol 2015;24(8):561-566.
4. Doddaballapur S. Microneedling with dermaroller. J Cutan AesthetSurg 2009;2:110-1.10
5. Aust MC, Reimers K, Kaplan HM, Stahl F, et al. Percutaneous collageninduction-regeneration in place of cicatrisation? J Plast Reconstr Aesthet Surg 2011;64:97-107.11.
6. Schwarz M, Laaff H. A prospective controlled assessment of microneedling with the Dermaroller device. Plast Reconstr Surg 2011;127:146e-148e.14.
7. Hou A, Cohen B, Haimovic A, Elbuluk N. Microneedling: A Comprehensive Review. Dermatol Surg. 2017 Mar;43(3):321-339

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion in the study if they are age 60 or older and have dermatoporosis of the dorsal forearms as defined by any or all of the following: white pseudoscars, senile purpura, or skin atrophy.

Exclusion Criteria:

* Exclusion criteria: Patients with liver disease, heart disease, active infection, keloid predisposition, immunosuppression, genetic predisposition to poor wound healing, active cancer in the treatment area, bleeding disorders, pregnancy or nursing, taking the medication isotretinoin, with open wounds, sores or irritated skin in the treatment area, allergy to stainless steel or anesthetics, or skin phototype 4 or greater will be excluded from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin thickness | one year
  Thickness of skin as measured by skin biopsy
Skin thickness ultrasound | 6 months
  Thickness of skin as measured by ultrasound

SECONDARY OUTCOMES:
Dermatology-related quality of life | six months and one year
  Dermatology quality of life index
Number of ecchymoses | six months and one year
  Number of ecchymoses

CONTACTS AND LOCATIONS:
Overall Officials: Richard M McLarney, MD, Principal Investigator — Resident

IPD SHARING:
Plan to Share IPD: No